CLINICAL TRIAL: NCT02950623
Title: Microbiological Comparative Study Between Single Maxillary Denture Fabricated From Rapid Heat Cured Resin and Conventional Acrylic Resin Modified by Titanium Dioxide Nanoparticles
Brief Title: Microbiological Study on Maxillary Complete Dentures of Two Different Materials
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed mabrouk abd Elmawla mahmoud, Principal Investigator, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Hozaifa
Record Dates: First submitted 2016-10-23; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Denture Stomatitis
MeSH Terms: conditions — Stomatitis, Denture

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patients take titanium dioxide denture (Experimental): patients will receive titanium dioxide denture (made from conventional acrylic resin modified by titanium dioxide nanoparticles ) for 1 month in the initial phase of the trial then in the later phase after one month they will receive( rapid heat cured acrylic resin)denture
  Interventions: Other: titanium dioxide denture; Other: rapid heat denture
- patients take rapid heat denture (Placebo Comparator): patients will receive rapid heat denture for 1 month in the initial phase of the trial then in the later phase patients will receive titanium dioxide denture (made from conventional acrylic resin modified by titanium dioxide nanoparticles )
  Interventions: Other: titanium dioxide denture; Other: rapid heat denture

INTERVENTIONS:
Other: titanium dioxide denture — patients will receive titanium dioxide denture (made from acrylic resin with titanium dioxide nanoparticles ) for 1 month in the initial phase then in the second phase after one month they will receive( rapid heat cured acrylic resin)denture according to the principle of crossover design
Other: rapid heat denture — patients will receive rapid heat denture for 1 month in the initial phase of the trial then in the later phase patients will receive titanium dioxide denture (made from conventional acrylic resin modified by titanium dioxide nanoparticles ) according to the principle of crossover design

SUMMARY:
Cross over design the investigator divide participants to two groups group (A) will receive rapid heat cured denture base material and group (b) will receive the acrylic denture modified by titanium dioxide nanoparticles and after washout period alternatively group (a) will receive the acrylic denture modified by titanium dioxide nanoparticles AND group (b) will receive rapid heat cured denture base material the investigator will take swaps from dentures to count the anaerobic bacteria.

DETAILED DESCRIPTION:
First the investigator will take primary impression, and pour it obtain primary cast, then will fabricate special tray an take secondary impression and obtain master cast after that duplication of master cast will be done the investigator will make cross over design.and divide participants to two groups group (A) will receive rapid heat cured denture base material and group (b) will receive the acrylic denture modified by titanium dioxide nanoparticle and after washout period alternatively group (a) will receive the acrylic denture modified by titanium dioxide nanoparticle AND group (b) will receive rapid heat cured denture base material the investigator will take swaps from the different dentures to count the anaerobic bacteria by (CFU).

ELIGIBILITY:
Inclusion Criteria:

1. Completely edentulous maxillary arch and partially dentate mandibular arch with adequate interarch space.
2. The edentulous ridges should be covered by firm healthy mucosa. 3-Angle class I maxillomandibular relation. 4-Healthy and cooperative patient

Exclusion Criteria:

1. Patients with bad habits as severe clenching or bruxism, drug or alcohol addiction, moderate or heavy smoking (greater than 10 cigarettes per day).
2. Previous history of radiotherapy or chemotherapy.
3. Any skeletal problem dictates surgical intervention

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Microbiological investigation: Count of anaerobic bacteria on the fitting surface of denture by (CFU) unit | 6 months
  Microbiological investigation: Count of anaerobic bacteria on the fitting surface of denture by (CFU) unit

IPD SHARING:
Plan to Share IPD: Undecided